CLINICAL TRIAL: NCT07329569
Title: Treatment of Severe Ocular Chemical Burns by Subconjunctival Injection of Allogeneic Mesenchymal Stem Cells: An Open-Label, Single-Arm, Multicenter Phase II Trial
Acronym: SYMBOLCLINICAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DGT_2025_2; 170641 (Other Grant/Funding Number: Programme Hospitalier de Recherche Clinique 2017)
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Chemical Burns; Ocular Burns
Keywords: severe chemical burns of the ocular surface; subconjunctival administration of allogeneic BM-MSCs
MeSH Terms: conditions — Burns, Chemical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subconjunctival injection of 1 mL with 5 million allogeneic BM-MSCs; one repeat within 21 days. (Experimental): Subconjunctival injection of a 1 mL suspension containing 5 million allogeneic BM-MSCs. A single injection or one repeat injection may be administered within 21 days if corneal epithelialization remains below 25%, as assessed by an expert clinician at the Adolphe de Rothschild Foundation Hospital, based on evaluation performed 7 to 10 days after the first injection.
  Interventions: Biological: Subconjunctival injection of 1 mL with 5 million allogeneic BM-MSCs; one repeat within 21 days.

INTERVENTIONS:
Biological: Subconjunctival injection of 1 mL with 5 million allogeneic BM-MSCs; one repeat within 21 days. — Subconjunctival injection of a 1 mL suspension containing 5 million allogeneic BM-MSCs. A single injection or one repeat injection may be administered within 21 days if corneal epithelialization remains below 25%, as assessed by an expert clinician at the Adolphe de Rothschild Foundation Hospital, based on evaluation performed 7 to 10 days after the first injection.

SUMMARY:
Severe chemical burns of the eye are serious injuries that can cause intense inflammation of the ocular surface and destroy limbal epithelial stem cells, which are essential for corneal healing. These injuries may lead to severe vision loss, blindness, or even loss of the eye despite standard medical and surgical treatments. Current therapies aim to control inflammation and promote healing, but outcomes remain poor in the most severe cases.

This Phase II clinical trial, called SYMBOL-Clinical, is designed to evaluate the safety and potential effectiveness of allogeneic bone marrow-derived mesenchymal stem cells (BM-MSCs) administered by subconjunctival injection in patients with severe ocular chemical burns (stage VI according to the Dua classification). Mesenchymal stem cells have shown anti-inflammatory and tissue-protective effects in preclinical studies, mainly through the release of paracrine factors that support healing.

This is an open-label, single-arm, multicenter study conducted in 13 centers in France and coordinated by the Adolphe de Rothschild Foundation Hospital. Adult patients (18 years or older) with a recent severe chemical burn of the ocular surface (within 15 days of injury) may be eligible to participate.

Participants will receive a subconjunctival injection of 5 million allogeneic BM-MSCs in the affected eye. A second injection may be administered within 21 days if corneal healing remains insufficient, as assessed by an expert ophthalmologist. All injections are performed under strict sterile conditions, with local anesthesia and conscious sedation when needed.

The primary objective of the study is to assess:

Safety, by monitoring the occurrence, type, and severity of adverse events.

Effectiveness, defined as preservation of the eye without corneal perforation at 6 months after the first injection.

Secondary objectives include evaluating corneal epithelial healing, limbal stem cell deficiency, conjunctival fibrosis, ocular surface inflammation, visual acuity, corneal thickness, the need for additional eye surgeries, and the use of local immunosuppressive treatments over a 12-month follow-up period.

Patients will be followed closely with regular ophthalmologic examinations, imaging (including anterior segment OCT), visual acuity testing, and safety assessments for up to 12 months after treatment. The total duration of participation for each patient is approximately 13 months, and the overall study duration is expected to be up to 49 months.

The study plans to enroll between 12 and 21 evaluable patients, using a two-stage Simon design to allow early stopping if the treatment does not show sufficient benefit.

The results of this study may help determine whether subconjunctival injection of allogeneic mesenchymal stem cells is a safe and promising treatment option for patients with the most severe forms of ocular chemical burns.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Unilateral or bilateral chemical burn of the ocular surface
* Severe ocular chemical burn of at least one eye, classified as stage VI according to the Dua severity classification (involving the entire limbus and conjunctiva)
* Time from chemical injury to enrollment ≤ 15 days
* Patient has received full study information and has provided written informed consent
* Affiliated with or beneficiary of a social security or health insurance system

Exclusion Criteria:

* Imminent corneal perforation (loss of more than two-thirds of corneal thickness)
* Ocular infection
* Eyelid tissue loss with permanent corneal exposure
* Known allergy or hypersensitivity to human albumin preparations
* History of total or partial limbal stem cell deficiency prior to the chemical injury
* Uncontrolled glaucoma prior to the ocular burn
* Recipient of a solid organ or cell transplant
* Severe or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, psychiatric, or cardiac disease, or any uncontrolled intercurrent illness
* Active infection, including chronic or localized infections
* History of malignancy (except completely resected localized basal cell carcinoma of the skin or cervical carcinoma in situ) within the past 5 years, whether treated or untreated, with or without evidence of recurrence or metastasis at screening
* Current treatment with systemic immunosuppressive medications (including systemic corticosteroids, TNF-α antagonists, azathioprine, methotrexate, mycophenolate mofetil)
* Adults under legal protection, individuals deprived of liberty by judicial or administrative decision, individuals receiving compulsory psychiatric care, or individuals admitted to a health or social care institution for purposes other than research
* Pregnant or breastfeeding women
* Women of childbearing potential who do not agree to use effective contraception throughout the study period (up to 12 months after the last injection)
* Participation in another interventional clinical trial during the study follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence, type, and severity of adverse events. | From the first allogeneic BM-MSC injection through 6 months after the first injection.
  incidence, type, and severity of adverse events.

SECONDARY OUTCOMES:
Efficacy: Absence of corneal perforation | 6 months after first injection of allogeneic BM-MSCs
  Absence of corneal perforation as assessed by the clinician; any suspected perforation will be confirmed by the coordinating expert physician based on slit-lamp photographs and corneal OCT images